CLINICAL TRIAL: NCT04867837
Title: Study of Four-factor Prothrombin Complex Concentrate, OCTAPLEX, in Patients With Acute Major Bleeding on Direct Oral Anticoagulant (DOAC) Therapy With Factor Xa Inhibitor
Brief Title: Study of OCTAPLEX in Patients With Acute Major Bleeding on DOAC Therapy With Factor Xa Inhibitor
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEX-210
Record Dates: First submitted 2021-04-19; First posted 2021-04-30 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Acute Major Bleeding
Keywords: Direct Oral Anticoagulant; Factor Xa Inhibitor
MeSH Terms: interventions — prothrombin complex concentrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Octaplex Low-dose (Experimental): Participants to receive 1 Octaplex infusion intravenously
  Interventions: Drug: Octaplex
- Octaplex High-dose (Experimental): Participants to receive 1 Octaplex infusion intravenously
  Interventions: Drug: Octaplex

INTERVENTIONS:
Drug: Octaplex — Four-factor prothrombin complex concentrate (4F-PCC)

SUMMARY:
This is a multicentre, prospective, randomised, double-blinded, group-sequential, parallel-group, adaptive design, phase 3 study to demonstrate the haemostatic efficacy and safety of four-factor prothrombin complex concentrate, OCTAPLEX, in patients with acute major bleeding on DOAC therapy with factor Xa inhibitor. Patients will be randomised 1:1 to either of two study groups: low-dose vs. high-dose OCTAPLEX.

ELIGIBILITY:
Inclusion Criteria:

1. Patients on oral factor Xa inhibitor therapy and with known or suspected baseline anti-factor Xa activity of at least 100 ng/mL:

   - Patients who received or who are believed by the investigator to have received a dose of oral factor Xa inhibitor and who have a baseline anti- factor Xa activity of at least 100 ng/mL according to the locally available test (e.g., chromogenic assay) performed outside of the study as part of standard of care

   OR
   * Patients who received or who are believed by the investigator to have received their latest dose of oral factor Xa inhibitor (e.g., rivaroxaban ≥10 mg, apixaban ≥2.5 mg, edoxaban ≥30 mg) ≤8 hours prior to enrolment

   OR

   -Patients who received or who are believed by the investigator to have received their latest dose of oral factor Xa inhibitor (e.g., rivaroxaban ≥10 mg, apixaban ≥2.5 mg, edoxaban ≥30 mg) >8 hours prior to enrolment or at an unknown time, but for whom the investigator suspects a baseline anti- factor Xa activity of at least 100 ng/mL and assesses that the administration of OCTAPLEX is clinically indicated
2. Aged ≥18 years
3. Patients who have given written informed consent or for whom written informed consent has been obtained from the patient's legally authorised representative on their behalf -Wherever possible, prospective written informed consent will be obtained before enrolment from the patient or, if they are incapable of providing it, from their legally authorised representative

   -If prospective written informed consent is not possible, deferred consent procedures will be permitted outside the US if approved by the local ethics committee or otherwise permitted under local regulations

   -When deferred consent procedures are used outside the US, written informed consent should be obtained from the patient as soon as they recover the capacity to provide it, or otherwise from their legally authorised representative
4. Patients who have acute major bleeding defined as follows:

   * Bleeding that is life-threatening or uncontrolled, e.g., with signs or symptoms of haemodynamic compromise, such as severe hypotension, poor skin perfusion, or low cardiac output that cannot be otherwise explained

OR

- Symptomatic bleeding in critical organs (intracranial, intraspinal, intraocular, gastrointestinal, retroperitoneal, intra-articular, pericardial, or intramuscular with compartment syndrome)

OR

- Acute overt bleeding associated with a fall in haemoglobin (Hgb) level of ≥2 g/dL, OR a Hgb level ≤8 g/dL if no baseline Hgb level is available, OR in the opinion of the investigator that the patient's Hgb level will fall to ≤8 g/dL with resuscitation

Exclusion Criteria:

1. Patients with 'Do not resuscitate' (DNR) orders
2. Patients with acute trauma for which reversal of DOAC therapy with factor Xa inhibitor alone would not be expected to control the bleeding event
3. Hgb decrease without accompanying evidence of source of bleeding
4. Acute coronary syndrome, ischaemic stroke or venous thromboembolism (VTE) within the preceding 3 months
5. Patients with a history, within the last 3 months, of disseminated intravascular coagulation (DIC) or hyperfibrinolysis
6. Patients with a known congenital bleeding disorder
7. Known inhibitors to coagulation factors II, VII, IX, or X; heparin-induced, type II thrombocytopenia; or immunoglobulin A (IgA) deficiency with known antibodies against IgA
8. Known hypersensitivity to plasma-derived products or heparin
9. Patients who received haemostatic agents, including plasma, platelets, PCC, activated PCC (aPCC), recombinant factor VIIa, or recombinant factor Xa inactivated-zhzo (andexanet alfa), for the current bleeding event prior to enrolment (antifibrinolytic drugs and local haemostatic agents are allowed)
10. Patients who received ticlopidine within 14 days, prasugrel within 7 days, ticagrelor within 5 days, dipyridamole within 1 day or cangrelor within 1 hour preceding the bleeding event
11. Patients on enoxaparin therapy for thromboembolic prophylaxis
12. A score of less than 7 on the Glasgow Coma Scale in non-intubated patients or an estimated intracerebral haematoma volume of more than 60 mL. (Patients intubated or sedated at the time of screening may be enrolled if intubation or sedation were done for non-neurologic reasons)
13. Patients with expected survival of less than 24 hours, in the opinion of the investigator (in collaboration with other medical experts as appropriate per usual local practice)
14. Patients scheduled to undergo surgery in less than 12 hours, with the exception of minor surgeries and invasive procedures which are allowed for diagnostic or therapeutic reasons or if intended to address a second (non-index) bleeding event
15. Patients who are pregnant or breastfeeding at the time of enrollment
16. Patients previously enrolled in this study
17. Patients participating in another interventional clinical treatment study currently or during the past 1 month prior to study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hemostatic efficacy | Within 24 hours after the start of initial management
  Binary outcome of effective (rating of excellent or good) or non-effective (rating of poor/none) in management of major bleeding events as assessed by the Independent Data Monitoring and Endpoint Adjudication Committee (IDMEAC) according to predefined criteria

SECONDARY OUTCOMES:
Change in endogenous thrombin potential (ETP) | From baseline to 1 hour after administration of drug
  Change in ETP as measured by thrombin generation assay
All-cause TEEs and All-cause Mortality | 30 days
  30-day event rate of thromboembolic events (TEEs) and all-cause mortality
Occurrence of Adverse Events (AEs) | From IMP infusion until Day 30
  Occurrence of any AEs from start of OCTAPLEX administration until end of study
Body Temperature | From day of IMP infusion until Day 30
  Temperature measured during a 48-hour follow-up period after OCTAPLEX administration and at discharge
Pulse | From day of IMP infusion until Day 30
  Pulse during a 48-hour follow-up period after OCTAPLEX administration and at discharge
Respiration rate | From day of IMP infusion until Day 30
  Respiration rate during a 48-hour follow-up period after OCTAPLEX administration and at discharge
Blood pressure | From day of IMP infusion until Day 30
  Blood pressure during a 48-hour follow-up period after OCTAPLEX administration and at discharge

OTHER OUTCOMES:
Change in Hgb | 48 hours after administration of drug
  Change in haematologic parameters based on complete blood count (CBC), i.e., Hgb, haematocrit (Hct), red blood cells (RBC), white blood cells (WBC), platelets, from baseline to 48 hours after OCTAPLEX administration
Change in haematocrit (Hct) | 48 hours after administration of drug
  Change in Hct from baseline to 48 hours after OCTAPLEX administration
Change in red blood cell (RBC) levels | 48 hours after administration of drug
  Change in RBC levels from baseline to 48 hours after OCTAPLEX administration
Change in white blood cell (WBC) levels | 48 hours after administration of drug
  Change in WBC levels from baseline to 48 hours after OCTAPLEX administration
Change in platelet levels | 48 hours after administration of drug
  Change in platelet levels from baseline to 48 hours after OCTAPLEX administration
Change in prothrombin time (PT) | 24 hours after administration of drug
  Change in prothrombin time from baseline during a 24-hour follow-up period after OCTAPLEX administration
Change in activated partial thromboplastin time (aPTT) | 24 hours after administration of drug
  Change in aPTT from baseline during a 24-hour follow-up period after OCTAPLEX administration
Change in Coagulation Parameters | 24 hour follow-up period
  Change in coagulation parameters (international normalised ratio [INR], prothrombin time [PT], activated partial thromboplastin time [aPTT], coagulation factors II, VII, IX, and X levels) from baseline during a 24-hour follow-up period after OCTAPLEX administration
Number of packed RBC concentrate (pRBC) transfusion | 48 hours after administration of drug
  The number of patients receiving one or more pRBC transfusions during a 48-hour follow-up period after OCTAPLEX administration.
Number of pRBC Units Transfused | 48-hour follow-up period
  The number of pRBC units transfused per patient during a 48-hour follow-up period after OCTAPLEX administration
Other Blood Products Used | 48-hour follow-up period
  The use of other blood products and/or haemostatic agents during a 48-hour follow-up period after OCTAPLEX administration
Use of Haemostatic Agents | 48 hours after administration of drug
  The use of haemostatic agents during a 48-hour follow-up period after OCTAPLEX administration.
Duration of Hospitalization | From admission to discharge, approximately 1-3 weeks
  Duration of hospitalization

CONTACTS AND LOCATIONS:
Locations (63):
- United States (10):
  - Harbor-UCLA Medical Center, Torrance, California
  - The University of Florida, Gainesville, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - OU Health - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Ascension Seton Medical Center Austin, Austin, Texas
  - Dell Seton Medical Center at the University of Texas, Austin, Texas
- Klinikum Klagenfurt am Wörthersee Anästhesiologie und Intensivmedizin, Klagenfurt, Austria
- Bosnia and Herzegovina (4):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - Univeristy Clinical Hospital Mostar, Mostar
  - Clinical Center University of Sarajevo, Sarajevo
  - University Clinical Center Tuzla, Tuzla
- Croatia (2):
  - Clinical Hospital Dubrava, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Centre Hospitalier Universitaire Francois Mitterand, Dijon, France
- Georgia (5):
  - Pineo Medical Ecosystem, Tbilisi
  - Tbilisi Institute of Medicine, Tbilisi
  - LTS ,, Israel-Geoargian Medical Research clinic Helsicore", Tbilisi
  - New Hospitals, Tbilisi
  - K.Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
- Germany (6):
  - Universitaetsklinikum Aachen, Klinik fuer Anaesthesiologie, Aachen
  - Universitatsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Essen, Klinik für Anästhesiologie und Intensivmedizin-Hufelandstraße, Essen
  - Universitaetsklinikum Frankfurt - Klinik fuer Anaesthesiologie, Intensivmedizin und Schmerztherapie, Frankfurt am Main
  - Heidelberg University Hospital Neurologische Universitätsklinik, Heidelberg
  - Universitatsklinikum Tubingen Hertie-lnstitut fur klinische Hirnforschung (HIH) / Neurologische Universitatsklinik, Tübingen
- Italy (6):
  - Ospedale Maggiore - IRCCS Istituto di Scienze Neurologiche di Bologna, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - San Raffaele Hospital, Milan
  - Azienda Ospedaliero -Universitaria di Modena, Modena
  - Ospedale Santa Maria della Misericordia, Perugia
  - Azienda Ospedaliero-Universitaria Senese, Siena
- Poland (4):
  - Ośrodek Badań Klinicznych BD Research, Iława
  - Clinical Research Center at Special Hospital Stefan Zeromski, Krakow
  - Military Institute of Medicine, Warsaw
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej w Łęcznej, Łęczna
- Spain (5):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Dr. Peset, Valencia
  - Hospital Universitario y Politecnico La Fe, Valencia
- Turkey (Türkiye) (10):
  - SBU Adana City Education and Research Hospital, Adana
  - Ankara University Faculty of Medicine, Ankara
  - İnönü University Faculty of Medicine, Battalgazi
  - Health Sciences University Bursa High Specialization Training and Research Hospital, Bursa
  - Istanbul University Istanbul Faculty of Medicine Department of Internal Diseases, Division of Hematology, Istanbul
  - Ege University Faculty of Medicine, Izmir
  - Kahramanmaraş Sütçü İmam University Faculty of Medicine, Kahramanmaraş
  - Mersin University Faculty of Medicine, Mersin
  - Ondokuz Mayıs University Faculty of Medicine, Samsun
  - Karadeniz Technical University, Trabzon
- Ukraine (6):
  - Public Non-profit Enterprise Clinical Emergency Care Hospital of Dnipro City Counsil, Dnipro
  - Public Non-profit Enterprise Regional Clinical Hospital of lvano-Frankivsk Regional Council, Ivano-Frankivsk
  - Public Non-profit Enterprise Central City Clinical Hospital of Ivano-Frankivsk City Council, Ivano-Frankivsk
  - Medical and Diagnostic Center of Private Enterprise of Private Manufacturing Company "Acinus", Kropyvnytskyi
  - Public Non-profit Enterprise Kyiv City Clinical Hospital #17 of Kyiv City Council Executive Body, Kyiv
  - Public Non-profit Enterprise of Lviv Regional Council Lviv Public non profit Regional Clinical Hospital, Lviv
- United Kingdom (3):
  - North Hampshire Hospitals NHS Foundation Trust, Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire
  - Nottingham University Hospital, Nottingham
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No